CLINICAL TRIAL: NCT03742986
Title: Phase II Trial of Nivolumab With Chemotherapy as Neoadjuvant Treatment in Inflammatory Breast Cancer (IBC)
Brief Title: Trial of Nivolumab With Chemotherapy as Neoadjuvant Treatment in Inflammatory Breast Cancer (IBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00890
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Nivolumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab; Paclitaxel; Doxorubicin; Cyclophosphamide; Docetaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HER2-negative, including TNBC or HR-positive (Experimental)
  Interventions: Drug: Nivolumab 360mg; Drug: Paclitaxel 80mg/m^2; Drug: Doxorubicin 60mg/m^2; Drug: Cyclophosphamide 600mg/m^2
- HER2-positive, independent of HR status (Experimental)
  Interventions: Drug: Nivolumab 360mg; Drug: Doxorubicin 60mg/m^2; Drug: Cyclophosphamide 600mg/m^2; Drug: Paclitaxel 80mg/m^2 or Docetaxel 75mg/m^2; Drug: Trastuzumab 8mg/kg and 6 mg/kg; Drug: Pertuzumab 840mg and 420mg

INTERVENTIONS:
Drug: Nivolumab 360mg — Nivolumab 360 mg IV on Day 1 of every 21 day cycle (Cycle 1-4)
Drug: Paclitaxel 80mg/m^2 — Paclitaxel 80mg/m^2 IV on Day of 1, 8, 15 of every 21 day cycle (Cycle 1-4)
  Arms: HER2-negative, including TNBC or HR-positive
Drug: Doxorubicin 60mg/m^2 — Doxorubicin 60 mg/m^2 IV on Day 1 of every 14 day cycle (Cycle 5-8)
Drug: Cyclophosphamide 600mg/m^2 — Cyclophosphamide 600mg/m^2 on Day 1 of every 14 day cycle (Cycle 5-8)
Drug: Paclitaxel 80mg/m^2 or Docetaxel 75mg/m^2 — Paclitaxel 80mg/m^2 on Day 1, 8, 15 of every 21 day cycle (Cycle 1-4) OR Docetaxel 75mg/m^2 on Day 1 of every 21 day cycle (Cycle 1-4)
  Arms: HER2-positive, independent of HR status
Drug: Trastuzumab 8mg/kg and 6 mg/kg — Trastuzumab 8mg/kg IV on Day 1 of Cycle 1 and then 6mg/kg IV on Day 1 of Cycle 2-4
  Arms: HER2-positive, independent of HR status
Drug: Pertuzumab 840mg and 420mg — Pertuzumab 840mg on Day 1 of Cycle 1 and then 420mg IV on Day 1 of Cycle 2-4
  Arms: HER2-positive, independent of HR status

SUMMARY:
Study of efficacy of nivolumab with neoadjuvant chemotherapy in patients with IBC

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the addition of nivolumab to chemotherapy improves pathologic complete response (pCR) in the breast and post-therapy lymph nodes evaluated histologically (ypT0/Tis ypN0) in patients with inflammatory breast cancer (IBC).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed inflammatory breast cancer without distant metastases and have not received prior chemotherapy or immunotherapy. All breast cancer subtypes are allowed: Triple negative breast cancer (TNBC); Hormone receptor (HR)-positive and human epidermal growth factor receptor 2 (HER2)-negative; HR-positive or HR-negative and HER2-positive

Exclusion Criteria:

* Clinical or radiologic evidence of distant metastases
* Malignancy that progressed within the last five years.
* Cardiac disease (history of and/or active disease)
* HIV positive
* Neuropathy ≥ Grade 2, per the NCI CTCAE v5.0
* Allogeneic stem cell or solid organ transplantation
* Autoimmune disease where in the opinion of the Investigator would preclude the use of immunotherapy
* Idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), or evidence of active pneumonitis
* Tuberculosis
* Pregnancy or lactation
* Treatment with CD137 agonists or immune checkpoint-blockade therapies, including anti-CD40, anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunosuppressive medications
* Cardiopulmonary dysfunction
* Clinically significant history of liver disease, including cirrhosis, autoimmune hepatic disorders, HIV infection, or active Hepatitis B or Hepatitis C
* Subject is pregnant or nursing
* Known hypersensitivity to the components of the study drugs(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryann Kwa, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Indiana University, Bloomington, Indiana
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be available as specified in publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HER2-negative, Including TNBC or HR-positive | HER2-positive, Independent of HR Status
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HER2-negative, Including TNBC or HR-positive | HER2-positive, Independent of HR Status | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 68.2 [52 to 75] | 49.75 [43 to 55] | 59 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Pathological Complete Response (pCR)
Description: pCR is defined as no histologic evidence of invasive tumor cells in the surgical breast specimen, axillary nodes, or sentinel node identified after neoadjuvant chemotherapy (ypT0/Tis ypN0).
Time Frame: up to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HER2-negative, Including TNBC or HR-positive | HER2-positive, Independent of HR Status
Number analyzed (Participants) | 4 | 4
Participants | 0 | 3

2. Primary Outcome: Number of Participants Who Had a Pathological Complete Response (pCR)
Description: as for outcome 1
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | HER2-negative, Including TNBC or HR-positive | HER2-positive, Independent of HR Status
Number analyzed (Participants) | 4 | 4
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | HER2-negative, Including TNBC or HR-positive | HER2-positive, Independent of HR Status
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-negative, Including TNBC or HR-positive (N=4) | HER2-positive, Independent of HR Status (N=4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Allergic Reaction (General disorders) | 0 | 1
Mediport Site Sepsis (Infections and infestations) | 0 | 1
Shortness of Breath (Dyspnea) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-negative, Including TNBC or HR-positive (N=4) | HER2-positive, Independent of HR Status (N=4)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Atrial Fibrilation (Cardiac disorders) | 4 | 1
Myocardial Infarction (Cardiac disorders) | 3 | 4
Palpitations (Cardiac disorders) | 3 | 3
Sinus Tachycardia (Cardiac disorders) | 4 | 3
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Colitis (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 3 | 3
Stomach Pain (Gastrointestinal disorders) | 4 | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 3 | 1
Allergic Reaction (General disorders) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 4 | 3
Aspartate Aminotransferase Increased (Investigations) | 3 | 2
Blood Bilirubin Increased (Investigations) | 4 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Chills (General disorders) | 3 | 3
Confusion (General disorders) | 4 | 3
Depression (Psychiatric disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 2
Dry Eye (Eye disorders) | 4 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 3
Dysgeusia (Nervous system disorders) | 3 | 2
Neutrophil Count Decreased (Investigations) | 2 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Platelet Count Decreased (Investigations) | 3 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Syncope (Nervous system disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 4 | 1
White Blood Cell Decreased (Investigations) | 2 | 3
Edema Face (General disorders) | 4 | 3
Edema Limbs (General disorders) | 2 | 3
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 4 | 2
Flatulence (Gastrointestinal disorders) | 4 | 3
Flushing (Vascular disorders) | 4 | 3
General Disorders and Administration Site Conditions (General disorders) | 3 | 4
Headache (Nervous system disorders) | 4 | 2
Hot Flashes (Vascular disorders) | 4 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 4
Hypotension (Vascular disorders) | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Infusion Related Reaction (General disorders) | 4 | 2
Lymphocyte Count Decreased (Investigations) | 2 | 2
Malaise (General disorders) | 3 | 4
Mucositis Oral (Gastrointestinal disorders) | 4 | 2
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Skin infection (Infections and infestations) | 2 | 4
Vaginal infection (Infections and infestations) | 3 | 4
Infections and Infestations (Infections and infestations) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Other Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 3 | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 2
Acute Kidney Injury (Renal and urinary disorders) | 4 | 3
Urinary Tract Infection (Renal and urinary disorders) | 3 | 4
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 4 | 3
Pruiritus (Skin and subcutaneous tissue disorders) | 3 | 4
Rash Acneiform (Skin and subcutaneous tissue disorders) | 4 | 3
Rash Maculo (Skin and subcutaneous tissue disorders) | 4 | 3
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 3 | 4
Folliculitis (Skin and subcutaneous tissue disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03742986/Prot_SAP_001.pdf